CLINICAL TRIAL: NCT03207048
Title: Repetitive Transcranial Magnetic Stimulation (rTMS) to Improve Cognitive Function and Prevent Relapses in Bipolar Patients
Brief Title: A Study of Repetitive Transcranial Magnetic Stimulation in Bipolar Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Psychiatric Hospital (Other Government)
Responsible Party: Principal Investigator, Kangguang Lin, Dr., Guangzhou Psychiatric Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Guangzhou Psychiatric Hospital
Record Dates: First submitted 2017-06-30; First posted 2017-07-02 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Cognitive Impairment; Relapse; Bipolar Disorder
MeSH Terms: conditions — Cognitive Dysfunction; Recurrence; Bipolar Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active rTMS (Experimental): 10 Hz repetitive transcranial magnetic stimulation (rTMS) applied to the left dorsolateral prefrontal cortex (L-DLPFC) for 15 mins each time, 5 times per week for up to 6 weeks (interrupt for 1-2 weeks after 10 times).
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Sham rTMS (Sham Comparator): Sham repetitive transcranial magnetic stimulation
  Interventions: Device: Sham repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — Daily left DLPFC, at 110% motor threshold, with a frequency of 10 Hz. Stimulation will be applied in 3-second trains with a 15-second inter-train interval, for 50 trains per session
  Arms: Active rTMS
Device: Sham repetitive transcranial magnetic stimulation — Sham Transcranial Magnetic Stimulation
  Arms: Sham rTMS

SUMMARY:
This study will investigate the effect of Repetitive transcranial magnetic stimulation (rTMS) on cognition and long-term clinical outcomes of bipolar patients.

DETAILED DESCRIPTION:
Cognitive deficits are core features of bipolar disorder. Preliminary evidence shows that repetitive transcranial magnetic stimulation (rTMS) might have positive effects in enhancing cognition and improving clinical symptoms in patients with depression. This study will investigate the effect of rTMS on cognition and long-term outcomes (12 month) of bipolar patients.

ELIGIBILITY:
Inclusion Criteria:

* Bipolar Type I or II subjects diagnosed according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-5)
* Age 18-60 years
* Rating on 24-items Hamilton Depression Rating Scale (HAMD)<18
* Rating on the Young Mania Rating Scale (YMRS) < 12

Exclusion Criteria:

* History of any DSM-IV Axis I diagnosis other than BD Type I or II
* Implanted medication pump or cardiac pacemaker;
* Have had prior brain surgery
* Any metal in the head (except in mouth)
* Any disease of increased Intracranial pressure
* Suicide attempt
* Pharmacotherapy
* unstable medical conditions
* in the process of changing and redrawing withdrawing psychoactive medications within the past 4 weeks (except for sleeping medications such as benzodiazepines)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Changes in the MATRICS Consensus Cognitive Battery | one weeks after the completion of the rTMS treatment)
  Changes in neurocognitive and social function (measured by the The MATRICS Consensus Cognitive Battery) after 2 session of rTMS treatments (20 times)

SECONDARY OUTCOMES:
relapses of depressive and/or hypo/mania episode | 12 months
  The number of patients who have depression and/or hyop/mania episodes over period of 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: kangguang Lin, MD; PhD, Principal Investigator — Guangzhou Brain hospital (Guangzhou Psychiatric Hospital)
Locations (1):
- Guangzhou Brain hospital(Guangzhou Huiai Hospital), Guangzhou, Guangdong, China

REFERENCES:
- [Background] Martin DM, McClintock SM, Forster JJ, Lo TY, Loo CK. Cognitive enhancing effects of rTMS administered to the prefrontal cortex in patients with depression: A systematic review and meta-analysis of individual task effects. Depress Anxiety. 2017 Nov;34(11):1029-1039. doi: 10.1002/da.22658. Epub 2017 May 24. PMID 28543994
- [Background] Kedzior KK, Schuchinsky M, Gerkensmeier I, Loo C. Challenges in comparing the acute cognitive outcomes of high-frequency repetitive transcranial magnetic stimulation (HF-rTMS) vs. electroconvulsive therapy (ECT) in major depression: A systematic review. J Psychiatr Res. 2017 Aug;91:14-17. doi: 10.1016/j.jpsychires.2017.03.002. Epub 2017 Mar 2. PMID 28288306